CLINICAL TRIAL: NCT01343056
Title: Program Reinforcement Impacts Self Management
Brief Title: Program Reinforcement Impacts Self Management (PRISM)
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Linda Siminerio, Linda Siminerio, RN, PhD, CDE, Executive Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO10090392
Record Dates: First submitted 2011-04-19; First posted 2011-04-27 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Self Management Education (DSME); Diabetes; Self Management Support (SMS)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Office Staff follow up education (Active Comparator): A designee in the office staff shall be assigned to follow up with the patient for for behavioral goal setting attainment. The office staff will call patients monthly to monitor goal attainment. It will be suggested that they phone the participant monthly but researchers will observe how and if they provide follow up.
  The intervention is the follow up goal attainment and office staff have been trained on elements of goal attainment.
  Interventions: Behavioral: Office Staff Support
- Peer follow up education (Active Comparator): A person with diabetes trained as a "peer" shall meet the participant at their 6 week follow up visit and then call the participant monthly to monitor behavioral goal attainment.The intervention is the follow up goal attainment and peers have been trained on elements of goal attainment.
  Interventions: Behavioral: Peer Support
- Usual Care (Active Comparator): ADA Recognition maintains the standard that a follow up to diabetes education must occur from 3-6 month post education. This one phone call will be made by the diabetes educator. The intervention is the diabetes educator making a phone call to the patient to ask how they are doing.
  Interventions: Behavioral: Usual Care Support
- Educator support follow up (Active Comparator): A diabetes educator will provide follow up support and make monthly call to the patient to ascertain behavioral goal setting attainment. The diabetes educator uses behavioral goal setting as an education intervention. The educator calls patient to determine goal attainment. That is the intervention.
  Interventions: Behavioral: Educator Support

INTERVENTIONS:
Behavioral: Office Staff Support — The intervention includes the Office staff of primary care practices trained to provide diabetes support for behavioral goal setting were tasked to follow up with patients via phone following completion of diabetes self-management education.
  Arms: Office Staff follow up education
Behavioral: Peer Support — Community peers trained to provide diabetes support for behavioral goal setting were tasked to follow up with patients via phone following completion of diabetes self-management education.
  Arms: Peer follow up education
Behavioral: Usual Care Support — Diabetes educators provided patient follow up for behavioral goal setting support according to traditional clinical guidelines following completion of diabetes self-management.
  Arms: Usual Care
Behavioral: Educator Support — Diabetes educators provided patient follow up for behavioral goal setting support that was problem-focused and patient centered.
  Arms: Educator support follow up

SUMMARY:
Patients who receive DSME (Diabetes Self Management Education) will be enrolled in a 4 arm, randomized study with each group receiving a different method of follow up. The 4 arms will be evaluated based on clinical indicators, goal achievement and patient satisfaction.

DETAILED DESCRIPTION:
As the diabetes burden worsens, the need for people to become more involved in self-management will increase. Research has demonstrated that diabetes self-management education (DSME) can improve HbA1C levels by 0.76%. While the rates of diabetes are increasing, the numbers of educators available are shrinking. This is a particular hardship in underserved and military communities where the supply of health care providers is already scarce. Our investigative team has led efforts in supporting DSME in the PA state-wide deployment of the Chronic Care Model (CCM) and reported findings nationally on innovative ways to increase the pool of education services by integrating educators into primary care, establishing nurse clinics in underserved communities and demonstrating that an educator position could be sustained by reimbursement. A 0.76% reduction associated to DSME can be considered an enormous benefit and is equivalent to the impact of most pharmacologic treatments for diabetes. Unfortunately, however the benefits of DSME decrease over time. This suggests that sustained improvements require contact and follow-up. SMS is defined as the process of ongoing support of patient self-care, to sustain the gains following DSME. There is often confusion among the terms self-management education (DSME) and self-management support (SMS). DSME is associated with the provision of knowledge and skills training delivered by a health care professional, e.g. nurses, dietitians, etc. SMS is defined as the process of making and refining changes in health care systems (and the community) to support patient self-care and maintain the gains made following DSME. We know that SMS is currently provided by diabetes educators, but only one 3-6 month follow up is usual care. It has been suggested that SMS can be provided by community workers, peers with diabetes, and office staff within community sites, like PCP offices, and wellness centers, etc. The National Standards for DSME and American Diabetes Association (ADA) Education Recognition Program (ERP) require that SMS approaches be delivered and documented, yet no evidence has been provided to define who should deliver it and how often. This uncertainty has led to many programs delivering SMS in an unstructured, non-standardized and at times haphazard fashion. Practical approaches designed for providing SMS have the potential to sustain improvements. The objective of this study is to compare Self-Management Support (SMS) interventions following Diabetes Self-Management Education (DSME) and determine which will be more likely to maintain improvements in behavioral and clinical outcomes following DSME while achieving patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* A person with diabetes referred for diabetes education

Exclusion Criteria:

* Gestational diabetes and pregnancy
* If a person has recently had diabetes education, they will not be enrolled in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Siminerio, RN, PhD, CDE, Principal Investigator — University of Pittsburgh; Robert Gabbay, MD, PhD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siminerio L, Ruppert KM, Gabbay RA. Who can provide diabetes self-management support in primary care? Findings from a randomized controlled trial. Diabetes Educ. 2013 Sep-Oct;39(5):705-13. doi: 10.1177/0145721713492570. Epub 2013 Jun 19. PMID 23782622

RESULTS

PARTICIPANT FLOW:
Groups:
- Office Staff Follow up of Diabetes Education: A designee in the office shall be assigned to follow up with the patient for goal attainment. It was suggested that they phone the participant monthly. Staff also received training on how best to provide support to patients.
- Peer Follow up of Diabetes Education: A person with diabetes trained as a "peer" met with the participant at their 6 week follow up visit and then called the participant monthly to monitor goal attainment.
- Usual Care: ADA Recognition maintains the standard that a follow up to diabetes education must occur from 3-6 month post education. This one phone call was made by a diabetes educator.
- Educator Support Follow up: A diabetes educator provided support to patients with periodic phone calls. Diabetes educators received training in ways to improve patient empowerment and best support their patients following diabetes education.
Period: Overall Study
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Started | 35 | 36 | 32 | 38
Completed | 28 | 31 | 29 | 29
Not Completed | 7 | 5 | 3 | 9
Not completed — Lost to Follow-up | 7 | 5 | 3 | 9

BASELINE CHARACTERISTICS:
Population: recruited type 2 diabetes patients who were referred for diabetes education
Groups:
- Office Staff Follow up of Diabetes Education: A designee in the office shall be assigned to follow up with the patient for goal attainment. It will be suggested that they phone the participant monthly but researchers will observe how and if they provide follow up.
  Four different methods of follow up of goal attainment post diabetes education shall be evaluated.: The four arms are described. All participants will receive a 6 week, 3 month and 6 month office visit where they will complete surveys and have blood work for HbA1C and Lipids.
- Peer Follow up of Diabetes Education: A person with diabetes trained as a "peer" shall meet the participant at their 6 week follow up visit and then call the participant monthly to monitor goal attainment.
  Four different methods of follow up of goal attainment post diabetes education shall be evaluated.: The four arms are described. All participants will receive a 6 week, 3 month and 6 month office visit where they will complete surveys and have blood work for HbA1C and Lipids.
- Usual Care: ADA Recognition maintains the standard that a follow up to diabetes education must occur from 3-6 month post education. This one phone call will be made by the diabetes educator.
  Four different methods of follow up of goal attainment post diabetes education shall be evaluated.: The four arms are described. All participants will receive a 6 week, 3 month and 6 month office visit where they will complete surveys and have blood work for HbA1C and Lipids.
- Educator Support Follow up: A diabetes educator will provide follow up support.
  Four different methods of follow up of goal attainment post diabetes education shall be evaluated.: The four arms are described. All participants will receive a 6 week, 3 month and 6 month office visit where they will complete surveys and have blood work for HbA1C and Lipids.
- Total: Total of all reporting groups
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up | Total
Number analyzed (Participants) | 35 | 36 | 32 | 38 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 32 | 38 | 141
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13.4) | 64 (10) | 60 (12) | 60 (10) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 16 | 20 | 80
  Male | 10 | 17 | 16 | 18 | 61
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 32 | 38 | 141

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C (HbA1C, %)
Time Frame: 6 months
Population: Number of participants analyzed represents the number of participants who completed a 6 month follow up visit and, therefore, differs from numbers reported in the Participant Flow Module.
Measure: Median (Full Range); unit: percentage of glycosolated hemoglobin
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 28 | 31 | 29 | 29
percentage of glycosolated hemoglobin | 6.8 [5.2 to 9.6] | 7.6 [5.4 to 11.6] | 6.8 [5.0 to 8.8] | 7.1 [5.9 to 10.2]

2. Secondary Outcome: Total Cholesterol (mg/dL)
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/dL
Groups:
- Office Staff Follow up Education: A designee in the office staff shall be assigned to follow up with the patient for goal attainment. The office staff will call patients monthly to monitor goal attainment. It will be suggested that they phone the participant monthly but researchers will observe how and if they provide follow up.
  Office Staff Support: Office staff of primary care practices trained to provide diabetes support were tasked to follow up with patients via phone following completion of diabetes self-management education.
- Peer Follow up Education: A person with diabetes trained as a "peer" shall meet the participant at their 6 week follow up visit and then call the participant monthly to monitor goal attainment.
  Peer Support: Community peers trained to provide diabetes support were tasked to follow up with patients via phone following completion of diabetes self-management education.
- Usual Care: ADA Recognition maintains the standard that a follow up to diabetes education must occur from 3-6 month post education. This one phone call will be made by the diabetes educator.
  Usual Care Support: Diabetes educators provided patient follow up support according to traditional clinical guidelines following completion of diabetes self-management.
- Educator Support Follow up: A diabetes educator will provide follow up support and make monthly call to the patient to ascertain goal attainment.
  Educator Support: Diabetes educators provided patient follow up support that was problem-focused and patient centered.
Arm/Group | Office Staff Follow up Education | Peer Follow up Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 28 | 31 | 29 | 29
mg/dL | 169 [100 to 205] | 159 [121 to 369] | 175 [129 to 321] | 150 [27 to 210]

3. Secondary Outcome: High Density Lipoprotein (HDL, mg/dL)
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 28 | 31 | 29 | 29
mg/dL | 46 [29 to 70] | 46 [35 to 67] | 39 [32 to 53] | 39 [23 to 84]

4. Secondary Outcome: Low Density Lipoprotein (LDL, mg/dL)
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 28 | 31 | 29 | 29
mg/dL | 86 [36 to 139] | 81 [59 to 274] | 103 [38 to 203] | 39 [23 to 84]

5. Secondary Outcome: Change in Diabetes Empowerment Scale- Short Form (DES-SF) Scores
Description: The DES-SF is a validated, 8 item scale that measures the self-efficacy of patients with diabetes. Responses are selected from a 5-point Likert scale (Strongly Disagree (1), Somewhat Disagree (2), Neutral (3), Somewhat Agree (4), Strongly Agree (5)). The scale is scored by averaging the scores of all completed items (sum of scores divided by 8).
  A positive number represents an improvement in overall patient self-efficacy (empowerment) from the baseline score and 6 month follow up time point.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 28 | 31 | 29 | 29
units on a scale | 3.9 (.8) | 4.1 (.7) | 4.0 (.9) | 4.5 (.4)

6. Secondary Outcome: Body Mass Index
Description: Body Mass Index is a weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters and used as an indicator of obesity and underweight.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: kg/m^2
Arm/Group | Office Staff Follow up Education | Peer Follow up Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 26 | 25 | 21 | 25
kg/m^2 | 35.1 [23.5 to 57] | 31.8 [23.2 to 47.1] | 32.3 [23.8 to 48] | 33.9 [24.9 to 50.2]

7. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure is the pressure when the heart is at rest between beats.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 26 | 25 | 21 | 26
mmHg | 78 [50 to 109] | 78 [60 to 92] | 78 [58 to 90] | 75 [60 to 92]

8. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure is the pressure when the heart beats while pumping blood.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Office Staff Follow up Education | Peer Follow up Education | Usual Care | Educator Support Follow up
Number analyzed (Participants) | 26 | 25 | 21 | 26
mmHg | 129 [108 to 155] | 130 [112 to 156] | 132 [102 to 150] | 132 [110 to 158]

ADVERSE EVENTS:
Arm/Group | Office Staff Follow up of Diabetes Education | Peer Follow up of Diabetes Education | Usual Care | Educator Support Follow up
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/32 | 0/38
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/32 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes